CLINICAL TRIAL: NCT04504799
Title: Validation of the New HAG-B19 Scale for Measuring Lean and Fat Body Masses by Comparison With Routinely Used Bioelectrical Impedance Analysis and Dual X-Ray Absorptiometry in Western Healthy Adults: The Geneva HAG-BIA Study
Brief Title: Validation of the New HAG-B19 Scale for Measuring Lean and Fat Body Masse
Acronym: HAG-BIA
Status: Completed | Type: Observational
Sponsor: Prof. Claude Pichard (Other)
Responsible Party: Sponsor-Investigator, Prof. Claude Pichard, Head, Clinical Nutrition, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2020-01613
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Body Composition
Keywords: Body composition; Bioimpendance analysis; Physical activity; Nutrition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Body composition measurement with HAG-BIA scale — Bio-impendance analysis

SUMMARY:
Body composition measurement is an important tool for assessing the physical condition of sick or healthy people, as well as for monitoring changes in body composition and physical performance during diet and/or training. Many people self-monitor their body composition using portable and inexpensive assessment tools, but most of them have not been tested for accuracy and precision.

This study aims to assess the accuracy and precision of a new portable impedancemeter scale to measure body composition in comparison with proven techniques, such as 4-electrode electrical bioimpedance analysis and dual X-ray absorptiometry.

DETAILED DESCRIPTION:
This is an observational, prospective, cross-sectional study to evaluate the accuracy and precision of the new HAG-B19 in healthy Western adults. A stratified sampling method is used to recruit a heterogeneous sample of 160 subjects, covering a wide range of ages and body compositions according to gender specific BMI distributions in the population. Volunteers who signed the informed consent form are included in the study. A financial compensation of 50.- CHF is given to each participant (100.- to the 16 participants subjected to the DEXA measurements).

The body composition of each subject (FM, LBM and FM%) is assessed with sequential measurements using 3 HAG-B19 and 3 Nutriguard-M® devices (Data Input, Germany). FM% values measured by HAG-B19 are compared to values by Nutriguard-M® to assess the accuracy and precision of HAG-B19 (main objective). Intra- and inter-device variability are obtained by comparing the 3 repeated measurements and the 3 HAG-B19 devices (secondary objective). In a subgroup of 16 individuals, the FM% values measured by HAG-B19 are compared to DEXA measurements (secondary objective). Pearson correlations and Bland-Altman graphs are performed to assess the agreement of the measurements between the devices and paired t-tests are used to determine if there is a bias between the devices. The significance of the statistical analysis is fixed at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

Healthy Caucasians/Hispanics adults who signed the informed consent form (healthy defined as no chronic disease, no hospitalisation for the last 6 months, no physical disability)

Exclusion Criteria:

* BMI <18.5 or ≥ 30 kg/m2
* No informed consent form signed
* Inability to understand the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Medication impacting fluid and electrolyte balance (diuretics or calcium channel blocker)
* Moderate to intense level physical activity 2-3 h before measurement
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Caucasians/Hispanics adults
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Accuracy of percent fat mass measurement | 6 months
  Comparison between HAG-B19 and Nutriguard-M measurement

SECONDARY OUTCOMES:
Intra- and inter-device variability of percent fat mass measurement | 6 months
  Comparison of measurements within and between three HAG-B19 devices.
Accuracy of percent fat mass measurement compared to gold standard | 6 months
  Comparison between HAG-B19 and DEXA in 10 percents of participants

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichard, Prof, Study Director — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Geneva 14, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamilton-James K, Collet TH, Pichard C, Genton L, Dupertuis YM. Precision and accuracy of bioelectrical impedance analysis devices in supine versus standing position with or without retractable handle in Caucasian subjects. Clin Nutr ESPEN. 2021 Oct;45:267-274. doi: 10.1016/j.clnesp.2021.08.010. Epub 2021 Sep 6. PMID 34620328